CLINICAL TRIAL: NCT06912204
Title: Predictive Value of the mNutric Score and Survival Analysis in Critically Ill Patients Hospitalised in the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Harun Tolga Duran, associate proffessor, Amasya University
Other Study IDs: htd
Record Dates: First submitted 2025-03-29; First posted 2025-04-04 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Intensive Care Medicine
Keywords: mturtic score; intensiva care; mortality

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- survived
- non-survived: Patients who did not survive after 28 days

SUMMARY:
Our study is an observational study and the follow-up hematological tests of patients in the intensive care unit will be recorded during their first admission. In this study, routinely checked blood parameters in patients will be interpreted and mnutric scores created together with their clinical features will be recorded. Routine blood tests will be performed during these records and no intervention will be made. Only an observational study will be conducted.

DETAILED DESCRIPTION:
Written informed consent was obtained from all participants or participants whose signature could not be obtained and included in the study. Between 1 December 2024 and 1 April 2025, 85 critically ill patients admitted to the anaesthesia intensive care unit of our hospital were included in the study. Patients aged 18 years and older who were admitted to the ICU and followed for more than 24 hours were included in the study. Patients younger than 18 years, pregnant women and patients with gastrointestinal motility disorders were excluded from the study. Patients' demographic characteristics, including age, sex, and comorbidities, were recorded at the time of initial admission. Haemoglobin (Hb), white blood cell (WBC), lymphocyte, platelet, aspartate aminotransferase (AST), alanine aminotransferase (ALT), C-reactive protein (CRP) and albumin levels were recorded during the first hospitalisation. Sequential Organ Failure Assessment Score 2 (SOFA 2) and Apache 2 score values were recorded. The 28-day follow-up of these patients was recorded. Patients who died within 28 days and patients who survived were grouped as survivors. The use of vasoactive drugs, renal replacement therapy, the need for mechanical ventilation and the length of stay in the intensive care unit of the groups were recorded during the follow-up period. The nutrition team placed a nasogastric catheter in all patients and started enteral nutrition at 25-30 kcal/kg in patients without contraindications.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old , Patients who have been hospitalized for more than 24 hours

Exclusion Criteria:

* under 18 years old, pregnancy patients, Patients hospitalized for less than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical care patients admitted to the intensive care unit and no deaths within 24 hours
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
primer | 28-day follow-up period
  It was aimed to investigate the mnutric scores of patients who survived and did not survive after 28 days of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University Training and Research Hospital, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
patient outcome data
Supporting Information: Study Protocol

REFERENCES:
- [Background] Grillo-Ardila CF, Tibavizco-Palacios D, Triana LC, Rugeles SJ, Vallejo-Ortega MT, Calderon-Franco CH, Ramirez-Mosquera JJ. Early Enteral Nutrition (within 48 h) for Patients with Sepsis or Septic Shock: A Systematic Review and Meta-Analysis. Nutrients. 2024 May 22;16(11):1560. doi: 10.3390/nu16111560. PMID 38892494